CLINICAL TRIAL: NCT01032460
Title: Comparison of Two Novel Indirect Laryngoscopes to the Macintosh Laryngoscope in Patients With Cervical Spine Immobilization.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Hospital Galway (Other)
Responsible Party: John G Laffey, National University of Ireland, Galway
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMAC-3
Record Dates: First submitted 2009-12-14; First posted 2009-12-15 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-07

CONDITIONS: Immobilization
Keywords: airway; airway device; cervical spine immobilisation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- macintosh (Active Comparator)
  Interventions: Device: intubate with the macintosh laryngoscope
- C-MAC (Active Comparator)
  Interventions: Device: intubate with the C-MAC laryngoscope
- Airtraq (Active Comparator)
  Interventions: Device: intubate with the Airtraq device

INTERVENTIONS:
Device: intubate with the macintosh laryngoscope — intubate with the macintosh laryngoscope
  Arms: macintosh
Device: intubate with the C-MAC laryngoscope — intubate with the C-MAC laryngoscope
  Arms: C-MAC
Device: intubate with the Airtraq device — intubate with the Airtraq device
  Arms: Airtraq

SUMMARY:
It is essential that anaesthetists successfully perform orotracheal intubation in scenarios in which intubation is potentially more difficult, such as where the neck is immobilized.

The Airtraq® Laryngoscope and the CMAC are new intubating devices. They are designed to provide a view of the glottis without alignment of the oral, pharyngeal and tracheal axes.

These devices may be especially effective in situations where intubation of the trachea is potentially difficult.

The efficacy of these devices in comparison to the traditional Macintosh laryngoscope in situations where the cervical spine is immobilized is not known.

The investigators aim to compare the performances of the Airtraq® Laryngoscope and the CMAC to that of the Macintosh laryngoscope, the gold standard device, in patients in which the cervical spine has been immobilized by means of a Manual in-line stabilization of the spine.

Hypothesis: The primary hypothesis is that, in the hands of experienced anaesthetists, time to intubation would be shorter using the indirect laryngoscopes, than using the Macintosh laryngoscope in simulated difficult laryngoscopy.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 - 3
* Aged 18 - 85 years
* Written informed Consent
* No relevant drug allergies
* Mallampatti 1 - 2.

Exclusion Criteria:

* Patients unable to cooperate with airway assessment (2)
* Patients with predicted difficult intubation

  * Mallampatti III or IV
  * Thyromental distance < 6cm
  * Mouth opening < 3.5 cm
  * Cervical spine disease
  * Anteriorly protruding incisors
  * Poor Dentition (2)
  * Tumours, polyps or foreign bodies in the upper airway (2)
  * Patients with documented difficult airways (2).
  * Patients with history of or risk factors for gastric regurgitation (i.e. require rapid sequence induction of anaesthesia)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Rate of successful placement of Tube in the Trachea a. Failed intubation defined as requiring greater than 60s or which resulted in Oesophageal Intubation. b. Successful intubation confirmed by an investigator. | immediately

SECONDARY OUTCOMES:
Duration of Intubation attempt (successful Attempts only) a. Absolute time taken to perform successful tracheal intubation b. Number of successful intubations completed within 30 seconds. | immediatley
Tracheal Intubation attempts. a. Overall number of attempts at Intubation. b. Number of successful intubations on first attempt | immediately
Laryngeal View Obtained a. Cormac and Lehane Grading of Best Laryngeal View b. POGO score | immediately
Intubation Difficulty Scale score | immediately
Need for and number of optimisation Manoeuvres to aid tracheal intubation | immediately

CONTACTS AND LOCATIONS:
Locations (1):
- Galway University Hospital, Galway, Galway, Ireland